CLINICAL TRIAL: NCT01386593
Title: Single-center, Randomized, Open-label, Two-way Crossover Study to Characterize Phenotyping Metrics of the "Basel" Cocktail After CYP Induction or Inhibition in Healthy Male Subjects
Brief Title: Pharmacokinetic Study to Characterize Phenotyping Metrics of the "Basel" Cocktail After CYP Induction or Inhibition
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: University Hospital, Basel, Switzerland (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None
Other Study IDs: EKBB-89/11; 2011 DR 1074 (Other: Swissmedic)
Record Dates: First submitted 2011-06-29; First posted 2011-07-01 (Estimated); Last update posted 2015-04-17 (Estimated); Status verified 2015-04

CONDITIONS: Metabolic Detoxication, Phase I
Keywords: Cytochrome; Phenotyping; Pharmacokinetics
MeSH Terms: interventions — Ciprofloxacin; Paroxetine; Rifampin

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (3):
- (A) Baseline (Other)
  Interventions: Drug: "Basel" Cocktail
- (B) Inhibition (Other)
  Interventions: Drug: Basel cocktail+(Fluconazole, Ciprofloxacin, Paroxetine)
- (C) Induction (Other)
  Interventions: Drug: Basel cocktail + Rifampicin

INTERVENTIONS:
Drug: Basel cocktail+(Fluconazole, Ciprofloxacin, Paroxetine)
  Arms: (B) Inhibition
Drug: "Basel" Cocktail
  Arms: (A) Baseline
Drug: Basel cocktail + Rifampicin
  Arms: (C) Induction

SUMMARY:
The purpose of this study is to assess how the pharmacokinetic profiles of each drug of a cocktail of six approved drugs (so-called "Basel cocktail") change when the cytochrome P450 system is inhibited or induced.

ELIGIBILITY:
Inclusion Criteria:

* Male aged between 18 and 35 years (inclusive) at screening.
* No clinically significant findings on the physical examination at screening.
* Body mass index (BMI) between 18 and 28 kg/m2 (inclusive) and body weight at least 50 kg at screening.
* Systolic blood pressure (SBP) 100-145 mmHg, diastolic blood pressure (DBP) 50-90 mmHg and heart rate (HR) 45-90 bpm (inclusive).
* 12-lead electrocardiogram (ECG) without clinically relevant abnormalities at screening.
* Hematology and clinical chemistry results not deviating from the normal range to a clinically relevant extent at screening.
* Ability to communicate well with the investigator and to understand and comply with the requirements of the study.

Exclusion Criteria:

* Known hypersensitivity to any excipients of the drug formulations.
* Treatment with another investigational drug within 30 days prior to screening.
* History or clinical evidence of alcoholism or drug abuse within the 3-year period prior to screening.
* Positive results from urine drug screen at screening.
* Excessive caffeine consumption, defined as >800 mg per day at screening*.
* African or Hispanic ethnicity.
* History or clinical evidence of any disease and/or existence of any surgical or medical condition, which might interfere with the absorption, distribution, metabolism or excretion of the study drugs, or which might increase the risk for toxicity.
* Smoking within the last 3 months prior to screening.
* Previous treatment with any prescribed or OTC medications (including herbal medicines such as St John's Wort) within 2 weeks prior to the intended start of study.
* Loss of 250 ml or more of blood within 3 months prior to screening.
* Any circumstances or conditions, which, in the opinion of the investigator, may affect full participation in the study or compliance with the protocol.
* Legal incapacity or limited legal capacity at screening.

Ages: 18 Years to 35 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 16 (Actual)
Dates: Start 2011-05; Primary Completion 2012-01 (Actual); Study Completion 2012-01 (Actual)

PRIMARY OUTCOMES:
Area under the plasma concentration versus time curve from timepoint 0 to 24 h (AUC24h) of the "Basel Cocktail" after inhibition with ciprofloxacin, fluconazole and paroxetine and after induction with rifampicin.

SECONDARY OUTCOMES:
Area under the plasma concentration versus time curve from timepoint 0 to infinity (AUC0-inf) of the "Basel Cocktail" after inhibition with ciprofloxacin, fluconazole and paroxetine and after induction with rifampicin.
Peak Plasma Concentration (Cmax) of the "Basel Cocktail" after inhibition with ciprofloxacin, fluconazole and paroxetine and after induction with rifampicin.
Peak Time (Tmax) of the "Basel Cocktail" in plasma after inhibition with ciprofloxacin, fluconazole and paroxetine and after induction with rifampicin.
Plasma Halflife (t1/2) in the elimination phase of the "Basel Cocktail" after inhibition with ciprofloxacin, fluconazole and paroxetine and after induction with rifampicin.
Area under the concentration in oral fluid versus time curve from timepoint 0 to 24 h (AUC24h) of the "Basel Cocktail" after inhibition with ciprofloxacin, fluconazole and paroxetine and after induction with rifampicin.
Area under the concentration in oral fluid versus time curve from timepoint 0 to infinity (AUC0-inf) of the "Basel Cocktail" after inhibition with ciprofloxacin, fluconazole and paroxetine and after induction with rifampicin.
Peak Concentration (Cmax) of the "Basel Cocktail" in oral fluid after inhibition with ciprofloxacin, fluconazole and paroxetine and after induction with rifampicin.
Peak Time (Tmax) of the "Basel Cocktail" in oral fluid after inhibition with ciprofloxacin, fluconazole and paroxetine and after induction with rifampicin.
Halflife (t1/2) in the elimination phase of the "Basel Cocktail" in oral fluid after inhibition with ciprofloxacin, fluconazole and paroxetine and after induction with rifampicin.
Area under the concentration in dried blood spots versus time curve from timepoint 0 to 24 h (AUC24h) of the "Basel Cocktail" after inhibition with ciprofloxacin, fluconazole and paroxetine and after induction with rifampicin.
Area under the concentration in dried blood spots versus time curve from timepoint 0 to infinity (AUC0-inf) of the "Basel Cocktail" after inhibition with ciprofloxacin, fluconazole and paroxetine and after induction with rifampicin.
Peak Concentration (Cmax) of the "Basel Cocktail" in dried blood spots after inhibition with ciprofloxacin, fluconazole and paroxetine and after induction with rifampicin.
Peak Time (Tmax) of the "Basel Cocktail" in dried blood spots after inhibition with ciprofloxacin, fluconazole and paroxetine and after induction with rifampicin.
Halflife (t1/2) in the elimination phase of the "Basel Cocktail" in dried blood spots after inhibition with ciprofloxacin, fluconazole and paroxetine and after induction with rifampicin.

CONTACTS AND LOCATIONS:
Overall Officials: Manuel Haschke, MD, Principal Investigator — University Hospital, Basel, Switzerland
Locations (1):
- Phase I Research Unit, University Hospital, Basel, Switzerland

REFERENCES:
- [Derived] Derungs A, Donzelli M, Berger B, Noppen C, Krahenbuhl S, Haschke M. Effects of Cytochrome P450 Inhibition and Induction on the Phenotyping Metrics of the Basel Cocktail: A Randomized Crossover Study. Clin Pharmacokinet. 2016 Jan;55(1):79-91. doi: 10.1007/s40262-015-0294-y. PMID 26123704